CLINICAL TRIAL: NCT02842086
Title: A Phase 3, Randomized, Double-blind Study to Evaluate the Safety and Efficacy of Emtricitabine and Tenofovir Alafenamide (F/TAF) Fixed-Dose Combination Once Daily for Pre-Exposure Prophylaxis in Men and Transgender Women Who Have Sex With Men and Are At Risk of HIV-1 Infection
Brief Title: Study to Evaluate the Safety and Efficacy of Emtricitabine and Tenofovir Alafenamide (F/TAF) Fixed-Dose Combination Once Daily for Pre-Exposure Prophylaxis in Men and Transgender Women Who Have Sex With Men and Are At Risk of HIV-1 Infection
Acronym: DISCOVER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-412-2055; 2022-501763-40 (Other: European Medicines Agency); 2016-001399-31 (EudraCT Number)
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Pre-Exposure Prophylaxis of HIV-1 Infection
MeSH Terms: interventions — emtricitabine tenofovir alafenamide; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- F/TAF (Experimental): F/TAF+ F/TDF placebo for at least 96 weeks
  Interventions: Drug: F/TAF; Drug: F/TDF Placebo
- F/TDF (Experimental): F/TDF+ F/TAF placebo for at least 96 weeks
  Interventions: Drug: F/TDF; Drug: F/TAF Placebo
- Open-label (Experimental): Once all participants have been on blinded treatment for at least 96 weeks, the study will be unblinded and participants will be offered the option to continue on open-label F/TAF treatment for 96 weeks.
  Interventions: Drug: F/TAF
- Open-Label Extension (Experimental): Participants who remain on study at Open-label Week 96 will have the option to continue on open-label F/TAF treatment in the Open-label extension phase for 408 weeks.
  Interventions: Drug: F/TAF

INTERVENTIONS:
Drug: F/TAF — 200/25 mg tablet administered orally once daily
  Other Names: Descovy®
  Arms: F/TAF; Open-Label Extension; Open-label
Drug: F/TDF — 200/300 mg tablet administered orally once daily
  Other Names: Truvada®
  Arms: F/TDF
Drug: F/TAF Placebo — Tablet administered orally once daily
  Arms: F/TDF
Drug: F/TDF Placebo — Tablet administered orally once daily
  Arms: F/TAF

SUMMARY:
The primary objective of this study is to assess the rates of HIV-1 infection in Men (MSM) and transgender women (TGW) who have sex with men and who are administered daily emtricitabine/tenofovir alafenamide (F/TAF) or emtricitabine/tenofovir disoproxil fumarate (F/TDF) with a minimum follow-up of 48 weeks and at least 50% of participants have 96 weeks of follow-up after randomization.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be at high risk of sexual acquisition of HIV
* HIV-1 negative status
* MSM and TGW (male at birth) who have at least one of the following:

  * condomless anal intercourse with at least two unique male partners in the past 12 weeks (partners must be either HIV-infected or of unknown HIV status)
  * documented history of syphilis in the past 24 weeks
  * documented history of rectal gonorrhea or chlamydia in the past 24 weeks
* Adequate renal function: estimated glomerular filtration rate ≥ 60 mL/min according to the Cockcroft-Gault formula
* Adequate liver and hematologic function:

  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN) and total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
  * Absolute neutrophil count ≥ 1000/mm^3; platelets ≥ 75,000/mm^3; hemoglobin ≥ 10 g/dL

Key Exclusion Criteria

* Grade 3 or Grade 4 proteinuria or glycosuria that is unexplained or not clinically manageable.

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men and Transgender Women
Enrollment: 5399 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2027-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (73):
- United States (41):
  - Beverly Hills, California
  - Los Angeles, California
  - Newport Beach, California
  - Oakland, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Torrance, California
  - Aurora, Colorado
  - Denver, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Ft. Pierce, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Berkley, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Las Vegas, Nevada
  - Somers Point, New Jersey
  - Santa Fe, New Mexico
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Huntersville, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Austria (2):
  - Graz
  - Vienna
- Canada (3):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec
- Denmark (4):
  - Hvidovre, Capital Region
  - Aarhus N, Central Jutland
  - Copenhagen, RegionH
  - Odense
- France (4):
  - Nice, Alpe Maritimes
  - Marseille, Provence-Alpes-Côte d'Azur Region
  - Paris, Provence-Alpes-Côte d'Azur Region
  - Paris
- Germany (3):
  - Munich, Bavaria
  - Berlin
  - Frankfurt
- Ireland (2):
  - Dublin, Dublin
  - Dublin
- Italy (2):
  - Milan
  - Roma
- Amsterdam, Netherlands
- Spain (4):
  - Badalona, Barcelona
  - Barcelona
  - Madrid
  - Vigo
- United Kingdom (7):
  - Soho, London
  - Whitechapel, London
  - Edinburgh, Scotland
  - Brighton, Sussex
  - Birmingham
  - London
  - Manchester

REFERENCES:
- [Result] Hare B. The Phase 3 DISCOVER Study: Daily F/TAF or F/TDF for HIV Preexposure Prophylaxis [Presentation]. Conference on Retroviruses and Opportunistic Infections (CROI); 2019 04-07 March; Seattle, WA.
- [Result] Mayer KH, Molina JM, Thompson MA, Anderson PL, Mounzer KC, De Wet JJ, DeJesus E, Jessen H, Grant RM, Ruane PJ, Wong P, Ebrahimi R, Zhong L, Mathias A, Callebaut C, Collins SE, Das M, McCallister S, Brainard DM, Brinson C, Clarke A, Coll P, Post FA, Hare CB. Emtricitabine and tenofovir alafenamide vs emtricitabine and tenofovir disoproxil fumarate for HIV pre-exposure prophylaxis (DISCOVER): primary results from a randomised, double-blind, multicentre, active-controlled, phase 3, non-inferiority trial. Lancet. 2020 Jul 25;396(10246):239-254. doi: 10.1016/S0140-6736(20)31065-5. PMID 32711800
- [Derived] Wohl DA, Spinner CD, Flamm J, Hare CB, Doblecki-Lewis S, Ruane PJ, Molina JM, Mills A, Brinson C, Ramgopal M, Clarke A, Crofoot G, Martorell C, Carter C, Cox S, Hojilla JC, Shao Y, Das M, Kintu A, Baeten JM, Grant RM, Mounzer K, Mayer K. HIV-1 infection kinetics, drug resistance, and long-term safety of pre-exposure prophylaxis with emtricitabine plus tenofovir alafenamide (DISCOVER): week 144 open-label extension of a randomised, controlled, phase 3 trial. Lancet HIV. 2024 Aug;11(8):e508-e521. doi: 10.1016/S2352-3018(24)00130-9. Epub 2024 Jul 14. PMID 39008999
- [Derived] Cespedes MS, Das M, Yager J, Prins M, Krznaric I, de Jong J, Xiao D, Shao Y, Wong P, Kintu A, Carter C, Hoornenborg E, Ruane P, Phoenix J, Younis I, Halperin J. Gender Affirming Hormones Do Not Affect the Exposure and Efficacy of F/TDF or F/TAF for HIV Preexposure Prophylaxis: A Subgroup Analysis from the DISCOVER Trial. Transgend Health. 2024 Jan 31;9(1):46-52. doi: 10.1089/trgh.2022.0048. eCollection 2024 Feb. PMID 38312459
- [Derived] Zivich PN, Cole SR, Edwards JK, Glidden DV, Das M, Shook-Sa BE, Shao Y, Mehrotra ML, Adimora AA, Eron JJ. HIV Prevention Among Men Who Have Sex With Men: Tenofovir Alafenamide Combination Preexposure Prophylaxis Versus Placebo. J Infect Dis. 2024 Apr 12;229(4):1123-1130. doi: 10.1093/infdis/jiad507. PMID 37969014
- [Derived] Ogbuagu O, Ruane PJ, Podzamczer D, Salazar LC, Henry K, Asmuth DM, Wohl D, Gilson R, Shao Y, Ebrahimi R, Cox S, Kintu A, Carter C, Das M, Baeten JM, Brainard DM, Whitlock G, Brunetta JM, Kronborg G, Spinner CD; DISCOVER study team. Long-term safety and efficacy of emtricitabine and tenofovir alafenamide vs emtricitabine and tenofovir disoproxil fumarate for HIV-1 pre-exposure prophylaxis: week 96 results from a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet HIV. 2021 Jul;8(7):e397-e407. doi: 10.1016/S2352-3018(21)00071-0. PMID 34197772
- [Derived] Glidden DV, Das M, Dunn DT, Ebrahimi R, Zhao Y, Stirrup OT, Baeten JM, Anderson PL. Using the adherence-efficacy relationship of emtricitabine and tenofovir disoproxil fumarate to calculate background hiv incidence: a secondary analysis of a randomized, controlled trial. J Int AIDS Soc. 2021 May;24(5):e25744. doi: 10.1002/jia2.25744. PMID 34021709
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-412-2055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Canada, and the European Union. The first participant was screened on 02 September 2016. The data cut date for the end of blinded treatment phase was 12 December 2019.
Pre-assignment Details: 5857 participants were screened.
Groups:
- Descovy (DVY): Blinded Phase: Descovy (DVY; emtricitabine/tenofovir alafenamide [F/TAF] 200/25 mg) fixed-dose combination (FDC) tablet plus placebo-to-match Truvada (TVD) (emtricitabine/tenofovir disoproxil fumarate [F/TDF] 200/300 mg) FDC tablet administered orally once daily for at least 96 weeks.
- Truvada (TVD): Blinded Phase: TVD (F/TDF 200/300 mg) FDC tablet plus placebo-to-match DVY (F/TAF 200/25 mg) FDC tablet administered orally once daily for at least 96 weeks.
Period: Overall Study
Arm/Group | Descovy (DVY) | Truvada (TVD)
Started | 2700 | 2699
Completed (Completed the Double Blind Phase) | 2156 | 2206
Not Completed | 544 | 493
Not completed — Randomized but Never Treated | 6 | 6
Not completed — Still in Double-Blind Phase | 7 | 3
Not completed — Adverse Event | 18 | 20
Not completed — Death | 3 | 3
Not completed — Investigator's Discretion | 9 | 13
Not completed — Non-Compliance with Study Drug | 9 | 8
Not completed — Protocol Violation | 8 | 4
Not completed — Withdrew Consent | 205 | 194
Not completed — Lost to Follow-up | 274 | 236
Not completed — HIV-1 Infection | 5 | 6

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug. Participants were grouped according to the treatment they actually received.
Groups:
- Descovy (DVY): Blinded Phase: DVY (F/TAF 200/25 mg) FDC tablet plus placebo-to-match TVD (F/TDF 200/300 mg) FDC tablet administered orally once daily for at least 96 weeks.
- Total: Total of all reporting groups
Arm/Group | Descovy (DVY) | Truvada (TVD) | Total
Number analyzed (Participants) | 2694 | 2693 | 5387
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10.6) | 36 (10.7) | 36 (10.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Transgender Women | 45 | 29 | 74
Sex: Female, Male [Count of Participants; unit: Participants] — Reported data indicates sex at birth.
  Participants
    Female | 0 | 0 | 0
    Male | 2694 | 2693 | 5387
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 12 | 14 | 26
  Race: Asian | 113 | 120 | 233
  Race: Black/Mixed Black | 240 | 234 | 474
  Race: Native Hawaiian or Pacific Islander | 17 | 23 | 40
  Race: White | 2264 | 2247 | 4511
  Race: Other (Nonblack) | 45 | 50 | 95
  Race: Not Permitted | 3 | 5 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 635 | 683 | 1318
  Ethnicity: Not Hispanic or Latino | 2058 | 2008 | 4066
  Ethnicity: Not Permitted | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 191 | 162 | 353
  Austria | 35 | 42 | 77
  Denmark | 98 | 104 | 202
  France | 18 | 14 | 32
  Germany | 187 | 183 | 370
  Ireland | 40 | 38 | 78
  Italy | 37 | 21 | 58
  Netherlands | 31 | 40 | 71
  Spain | 219 | 195 | 414
  United Kingdom | 247 | 265 | 512
  United States | 1591 | 1629 | 3220
Hip Bone Mineral Density (BMD) [Mean (Standard Deviation); unit: g/cm^2] — Population: Hip Dual-Energy X-ray Absorptiometry (DXA) Analysis Set included all DXA substudy participants who were randomized and received at least one dose of study drug, and had nonmissing hip BMD value for the baseline visit. Participants were grouped according to the treatment they actually received.
  g/cm^2
    number analyzed (Participants) | 191 | 185 | 376
    (all) | 1.030 (0.1553) | 1.021 (0.1322) | 1.025 (0.1443)
Spine BMD [Mean (Standard Deviation); unit: g/cm^2] — Population: Spine DXA Analysis Set included all DXA substudy participants who were randomized and received at least one dose of study drug, and had nonmissing spine BMD value for the baseline visit. Participants were grouped according to the treatment they actually received.
  g/cm^2
    number analyzed (Participants) | 191 | 188 | 379
    (all) | 1.134 (0.1646) | 1.131 (0.1381) | 1.132 (0.1518)
Urine Beta-2 Microglobulin to Creatinine Ratio [Mean (Standard Deviation); unit: µg/g] — Population: Participants in Safety Analysis Set with available data were analyzed.
  µg/g
    number analyzed (Participants) | 2677 | 2676 | 5353
    (all) | 204.3 (951.77) | 188.5 (1010.19) | 196.4 (981.35)
Urine Retinol Binding Protein (RBP) to Creatinine Ratio [Mean (Standard Deviation); unit: µg/g] — Population: Participants in Safety Analysis Set with available data were analyzed.
  µg/g
    number analyzed (Participants) | 2686 | 2686 | 5372
    (all) | 148.8 (553.54) | 142.8 (256.64) | 145.8 (431.41)
Urine Protein (UP) and Urine Protein to Creatinine Ratio (UPCR) Categories [Count of Participants; unit: Participants] — The UPCR was only calculated when corresponding urine protein (UP) ≥ 4.0 mg/dL. The UPCR "≤ 200 mg/g" category includes both participants with UP < 4.0 mg/dL and participants with UPCR ≤ 200 mg/g. Population: Participants in Safety Analysis Set with available data were analyzed.
  Participants
    number analyzed (Participants) | 2687 | 2682 | 5369
    ≤ 200 mg/g | 2662 | 2657 | 5319
    > 200 mg/g | 25 | 25 | 50
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.96 (0.146) | 0.96 (0.148) | 0.96 (0.147)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of HIV-1 Infection Per 100 Person Years (PY)
Description: The incidence of HIV-1 infection rate per 100 PY was calculated as the number of participants who became HIV infected during the study after the first dose of study drug divided by the sum of all participants' years (where a year is 365.25 days) of follow-up while at risk of HIV infection during the study.
  HIV-1 infection is defined by one or more of the following criteria of contributing HIV tests performed via central lab or local lab:
  * Serologic evidence of seroconversion (reactive screening HIV Antigen/Antibody or Antibody test, confirmed by reactive HIV-1/HIV-2 differentiation assay), excluding HIV vaccinated participants, or
  * Virologic evidence of HIV-1 infection (positive qualitative HIV-1 RNA test or any detectable quantitative HIV-1 RNA test), or
  * Evidence of acute HIV-1 infection (reactive p24 Antigen or positive qualitative or quantitative RNA, in the absence of reactive HIV-1 Antibody results)
Time Frame: When all participants completed minimum follow-up of 48 weeks and at least 50% of the participants completed 96 weeks of follow-up after randomization or permanently discontinued from the study (maximum 125 weeks)
Population: The Full Analysis Set included all participants who were randomized into the study, received at least 1 dose of study drug, were not HIV positive on Day 1, and had at least 1 postbaseline HIV laboratory assessment.
Measure: Number (95% Confidence Interval); unit: HIV-1 infections per 100 PY
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2670 | 2665
HIV-1 infections per 100 PY | 0.160 [0.064 to 0.330] | 0.342 [0.191 to 0.564]
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Noninferiority was assessed using a 95.003% confidence interval (CI) constructed using a generalized model associated with a Poisson distribution and logarithmic link with the treatment group being the main effect and with a noninferiority margin of 1.62; Test type: Non-Inferiority — Noninferiority of DVY to TVD was to be concluded if the upper bound of the 2-sided 95.003% CI of the rate ratio (DVY group over TVD group) in the HIV infection incidence rate was less than 1.62; Rate Ratio = 0.468, 95.003% CI 2-sided [0.191 to 1.149]

2. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48 in the Blinded Phase
Description: Percent Change = Change from baseline at Week 48 visit/value at baseline * 100%.
Time Frame: Baseline, Week 48
Population: Hip Dual-Energy X-ray Absorptiometry (DXA) Analysis Set included all DXA substudy participants who were randomized and received at least one dose of study drug, and had nonmissing hip BMD value for the baseline visit. Participants were grouped according to the treatment they actually received. Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 159 | 157
Percent Change | 0.218 (2.3668) | -0.968 (2.4343)
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Hip BMD results were compared between the 2 treatment groups using analysis of variance (ANOVA), which included baseline TVD for pre-exposure prophylaxis (PrEP) and treatment as fixed effects; Test type: Superiority; p < 0.0001, ANOVA; Difference in least squares mean (LSM) = 1.142, 95% CI 2-sided [0.628 to 1.655]

3. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48 in the Blinded Phase
Description: Percent Change = Change from baseline at Week 48 visit/value at baseline * 100%.
Time Frame: Baseline, Week 48
Population: Spine DXA Analysis Set included all DXA substudy participants who were randomized and received at least one dose of study drug, and had nonmissing spine BMD value for the baseline visit. Participants were grouped according to the treatment they actually received. Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 160 | 159
Percent Change | 0.512 (2.9854) | -1.061 (2.9382)
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Spine BMD results were compared between the 2 treatment groups using ANOVA, which included baseline TVD for PrEP and treatment as fixed effects; Test type: Superiority; p < 0.0001, ANOVA; Difference in LSM = 1.567, 95% CI 2-sided [0.913 to 2.220]

4. Secondary Outcome: Percent Change From Baseline in Urine Beta-2-Microglobulin to Creatinine Ratio at Week 48 in the Blinded Phase
Description: Percent Change = Change from baseline at Week 48 visit/value at baseline * 100%.
  For urine creatinine, value of < 1 was handled as a missing value in its summary and the calculation of related ratios.
Time Frame: Baseline, Week 48
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug. Participants were grouped according to the treatment they actually received. Participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2346 | 2337
Percent Change | -10.6 [-42.0 to 25.9] | 15.4 [-22.9 to 97.2]
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Test type: Superiority; p < 0.0001, Van Elteren test — P-values were from the Van Elteren test stratified by baseline TVD for PrEP

5. Secondary Outcome: Percent Change From Baseline in Urine Retinol Binding Protein (RBP) to Creatinine Ratio at Week 48 in the Blinded Phase
Description: as for outcome 4
Time Frame: Baseline, Week 48
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2360 | 2354
Percent Change | 0.1 [-24.9 to 35.3] | 20.0 [-13.0 to 68.2]
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Test type: Superiority; p < 0.0001, Van Elteren test — P-values were from the Van Elteren test stratified by baseline TVD for PrEP

6. Secondary Outcome: Number of Participants by Urine Protein (UP) and Urine Protein to Creatinine Ratio (UPCR) Categories at Week 48 in the Blinded Phase
Description: The UPCR was only calculated when corresponding UP ≥ 4.0 mg/dL. The UPCR "≤ 200 mg/g" category includes both participants with UP < 4.0 mg/dL and participants with UPCR ≤ 200 mg/g.
Time Frame: Baseline, Week 48
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2355 | 2348
Participants
  ≤ 200 mg/g at Baseline; ≤ 200 mg/g at Week 48 | 2318 | 2295
  ≤ 200 mg/g at Baseline; > 200 mg/g at Week 48 | 16 | 35
  > 200 mg/g at Baseline; ≤ 200 mg/g at Week 48 | 12 | 8
  > 200 mg/g at Baseline; > 200 mg/g at Week 48 | 9 | 10
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Test type: Superiority; p = 0.0048, Rank analysis of covariance — P-value for difference between treatment groups in distributions of UPCR ≤ 200 mg/g versus > 200 mg/g was from the rank analysis of covariance adjusting for baseline category and baseline TVD for PrEP

7. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 48 in the Blinded Phase
Time Frame: Baseline, Week 48
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2370 | 2368
mg/dL | -0.01 (0.107) | 0.01 (0.111)
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Results were compared between the 2 treatment groups using the analysis of covariance (ANCOVA) model including baseline TVD for PrEP and treatment as fixed effects and baseline serum creatinine as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LSM = -0.02, 95% CI 2-sided [-0.02 to -0.01]

8. Secondary Outcome: Incidence of HIV-1 Infection Per 100 PY
Description: as for outcome 1
Time Frame: When all participants have 96 weeks of follow-up after randomization or permanently discontinued from the study (maximum 157 weeks)
Population: Participants in Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: HIV-1 infections per 100 PY
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2670 | 2665
HIV-1 infections per 100 PY | 0.159 [0.069 to 0.313] | 0.297 [0.166 to 0.490]
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Noninferiority was assessed using a 95.003% CI constructed using a generalized model associated with a Poisson distribution and logarithmic link with the treatment group being the main effect and with a noninferiority margin of 1.62; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Rate Ratio = 0.536, 95.003% CI 2-sided [0.227 to 1.264]

9. Secondary Outcome: Percent Change From Baseline in Hip BMD at Week 96 in the Blinded Phase
Description: Percent Change = Change from baseline at Week 96 visit/value at baseline * 100%.
Time Frame: Baseline, Week 96
Population: Participants in Hip DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 144 | 138
Percent Change | 0.565 (2.9379) | -1.048 (2.9277)
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Hip BMD results were compared between the 2 treatment groups using ANOVA, which included baseline TVD for PrEP and treatment as fixed effects; Test type: Superiority; p < 0.0001, ANOVA; Difference in LSM = 1.567, 95% CI 2-sided [0.896 to 2.237]

10. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 96 in the Blinded Phase
Description: Percent Change = Change from baseline at Week 96 visit/value at baseline * 100%.
Time Frame: Baseline, Week 96
Population: Participants in Spine DXA Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 145 | 142
Percent Change | 0.831 (3.4608) | -1.426 (3.5508)
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Difference in LSM = 2.253, 95% CI 2-sided [1.437 to 3.069]

11. Secondary Outcome: Percent Change From Baseline in Urine Beta-2-Microglobulin to Creatinine Ratio at Week 96 in the Blinded Phase
Description: Percent Change = Change from baseline at Week 96 visit/value at baseline * 100%.
  For urine creatinine, value of < 1 was handled as a missing value in its summary and the calculation of related ratios.
Time Frame: Baseline, Week 96
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2169 | 2195
Percent Change | -14.5 [-45.4 to 23.9] | 14.1 [-26.2 to 99.5]
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Test type: Superiority; p < 0.0001, Van Elteren test — P-values were from the Van Elteren test stratified by baseline TVD for PrEP

12. Secondary Outcome: Percent Change From Baseline in Urine RBP to Creatinine Ratio at Week 96 in the Blinded Phase
Description: as for outcome 11
Time Frame: Baseline, Week 96
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2188 | 2211
Percent Change | 0.3 [-27.1 to 35.7] | 21.4 [-13.8 to 73.9]
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Test type: Superiority; p < 0.0001, Van Elteren test — P-values were from the Van Elteren test stratified by baseline TVD for PrEP

13. Secondary Outcome: Number of Participants by UP and UPCR Categories at Week 96 in the Blinded Phase
Description: as for outcome 6
Time Frame: Baseline, Week 96
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2175 | 2199
Participants
  ≤ 200 mg/g at Baseline; ≤ 200 mg/g at Week 96 | 2134 | 2153
  ≤ 200 mg/g at Baseline; > 200 mg/g at Week 96 | 21 | 28
  > 200 mg/g at Baseline; ≤ 200 mg/g at Week 96 | 14 | 10
  > 200 mg/g at Baseline; > 200 mg/g at Week 96 | 6 | 8
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Test type: Superiority; p = 0.2163, Rank analysis of covariance — [p-value comment as in outcome 6, analysis 1]

14. Secondary Outcome: Change From Baseline in Serum Creatinine at Week 96 in the Blinded Phase
Time Frame: Baseline, Week 96
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2194 | 2218
mg/dL | 0.01 (0.114) | 0.03 (0.117)
Statistical Analysis 1: Comparison: Descovy (DVY) vs Truvada (TVD); Results were compared between the 2 treatment groups using the ANCOVA model including baseline TVD for PrEP and treatment as fixed effects and baseline serum creatinine as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LSM = -0.02, 95% CI 2-sided [-0.02 to -0.01]

15. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Time Frame: First dose date up to the data cut for end of blinded treatment (maximum: 157 weeks)
Population: Participants in Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2694 | 2693
percentage of participants | 93.7 | 93.6

16. Secondary Outcome: Percentage of Participants Experiencing Any Treatment-Emergent Laboratory Abnormality
Time Frame: First dose date up to the data cut for end of blinded treatment (maximum: 157 weeks)
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Descovy (DVY) | Truvada (TVD)
Number analyzed (Participants) | 2672 | 2665
percentage of participants | 76.1 | 79.1

ADVERSE EVENTS:
Time Frame: First dose date up to the data cut for end of blinded treatment (maximum: 157 weeks)
Description: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug. Participants were grouped according to the treatment they actually received.
Groups:
- Descovy (DVY): DVY (F/TAF 200/25 mg) FDC tablet plus placebo-to-match TVD (F/TDF 200/300 mg) FDC tablet administered orally once daily for at least 96 weeks.
- Truvada (TVD): TVD (F/TDF 200/300 mg) FDC tablet plus placebo-to-match DVY (F/TAF 200/25 mg) FDC tablet administered orally once daily for at least 96 weeks.
Arm/Group | Descovy (DVY) | Truvada (TVD)
All-Cause Mortality (participants affected / at risk) | 3/2694 | 3/2693
Serious Adverse Events (participants affected / at risk) | 202/2694 | 186/2693
Other Adverse Events (participants affected / at risk) | 2258/2694 | 2229/2693
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Descovy (DVY) (N=2694) | Truvada (TVD) (N=2693)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 7
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac flutter (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 3
Myocarditis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Pectus excavatum (Congenital, familial and genetic disorders) | 0 | 1
Sickle cell disease (Congenital, familial and genetic disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 2 | 0
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0
Ocular myasthenia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Enlarged uvula (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 2
Mesenteritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal rupture (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Proctitis (Gastrointestinal disorders) | 1 | 1
Rectal lesion (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 2 | 4
Death (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Sudden death (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Treatment failure (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Amyloidosis (Immune system disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 2 | 0
Abscess oral (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 2 | 3
Appendicitis (Infections and infestations) | 9 | 10
Appendicitis perforated (Infections and infestations) | 0 | 1
Brain abscess (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 7 | 5
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 1
Chronic tonsillitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 3 | 3
Endocarditis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Eye infection gonococcal (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 4
Gastroenteritis Escherichia coli (Infections and infestations) | 1 | 0
Gastroenteritis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis shigella (Infections and infestations) | 2 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Giardiasis (Infections and infestations) | 1 | 0
Gonorrhoea (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 2
Hepatitis A (Infections and infestations) | 6 | 2
Infected bite (Infections and infestations) | 1 | 1
Infective tenosynovitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 1
Large intestine infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lymphogranuloma venereum (Infections and infestations) | 1 | 1
Malaria (Infections and infestations) | 0 | 1
Measles (Infections and infestations) | 0 | 1
Meningitis streptococcal (Infections and infestations) | 1 | 0
Neurosyphilis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 1 | 1
Parotid abscess (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pharyngeal abscess (Infections and infestations) | 1 | 0
Plasmodium falciparum infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 4
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Proctitis chlamydial (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 3 | 1
Septic shock (Infections and infestations) | 1 | 1
Shigella infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 2
Tooth infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Viral pericarditis (Infections and infestations) | 0 | 1
Viral rash (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 2
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 4 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2
Reactive gastropathy (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 4 | 1
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 2
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Scan myocardial perfusion abnormal (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Facial paralysis (Nervous system disorders) | 1 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 1
Myelitis transverse (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Device dislocation (Product Issues) | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1
Alcohol use disorder (Psychiatric disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Delusion (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 5 | 3
Intentional self-injury (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 2 | 0
Personality disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 2 | 3
Schizoaffective disorder (Psychiatric disorders) | 0 | 1
Substance abuse (Psychiatric disorders) | 2 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 8 | 5
Suicide attempt (Psychiatric disorders) | 5 | 1
Acute kidney injury (Renal and urinary disorders) | 7 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal infarct (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 2
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Alcohol use (Social circumstances) | 1 | 0
Ligament operation (Surgical and medical procedures) | 0 | 1
Medical device removal (Surgical and medical procedures) | 0 | 1
Spinal fusion surgery (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Descovy (DVY) (N=2694) | Truvada (TVD) (N=2693)
Diarrhoea (Gastrointestinal disorders) | 479 | 451
Nausea (Gastrointestinal disorders) | 209 | 204
Fatigue (General disorders) | 180 | 181
Anal chlamydia infection (Infections and infestations) | 890 | 902
Gastroenteritis (Infections and infestations) | 171 | 141
Influenza (Infections and infestations) | 145 | 143
Nasopharyngitis (Infections and infestations) | 399 | 402
Oropharyngeal gonococcal infection (Infections and infestations) | 871 | 838
Pharyngeal chlamydia infection (Infections and infestations) | 215 | 186
Pharyngitis (Infections and infestations) | 166 | 108
Proctitis gonococcal (Infections and infestations) | 805 | 797
Syphilis (Infections and infestations) | 413 | 392
Upper respiratory tract infection (Infections and infestations) | 402 | 346
Urethritis (Infections and infestations) | 193 | 189
Urethritis chlamydial (Infections and infestations) | 346 | 314
Urethritis gonococcal (Infections and infestations) | 259 | 255
Exposure to communicable disease (Injury, poisoning and procedural complications) | 554 | 548
Headache (Nervous system disorders) | 206 | 209
Cough (Respiratory, thoracic and mediastinal disorders) | 152 | 136
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 172 | 165
Rash (Skin and subcutaneous tissue disorders) | 136 | 122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT02842086/Prot_003.pdf
  • Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT02842086/SAP_002.pdf